CLINICAL TRIAL: NCT07340294
Title: ClinicAL outComes of IntraVascular Lithotripsy Combined With Conventional Lesion Preparation in Patients With Moderate to Severe Coronary Artery Calcification
Acronym: CALC-IVL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Hospital of China Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); The People's Hospital of Liaoning Province (Other); Tianjin Forth Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0812
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Calcification; Calcific Coronary Arteriosclerosis
Keywords: atherosclerosi; calcification; coronary artery calcification
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Preconditioning Group (Experimental): Routine preconditioning strategy + IVL Routine Preconditioning Strategy plus IVL (IVL may be performed before, during, or after the routine preconditioning strategy, with IVL being mandatory).The ratio of the IVL catheter size to the reference vessel diameter of the target lesion is 1:1. The IVL catheter is inflated to 4 atmospheres (atm) at the target lesion and delivers 10 pulses, followed by deflation to restore blood perfusion. A maximum of 80 pulses may be delivered, and the IVL catheter can be repositioned within the lesion. For diffuse lesions involving different reference diameters, IVL catheters of different sizes may be utilized.
  Interventions: Device: Intensive Preconditioning Group
- Control group (Other): Routine preconditioning strategy This includes compliant balloons, non-compliant balloons, cutting/scoring balloons, excimer laser, and rotational atherectomy, to be determined at the operator's discretion.
  Interventions: Device: Routine preconditioning strategy

INTERVENTIONS:
Device: Intensive Preconditioning Group — Routine Preconditioning Strategy plus IVL (IVL may be performed before, during, or after the routine preconditioning strategy, with IVL being mandatory).The ratio of the IVL catheter size to the reference vessel diameter of the target lesion is 1:1. The IVL catheter is inflated to 4 atmospheres (atm) at the target lesion and delivers 10 pulses, followed by deflation to restore blood perfusion. A maximum of 80 pulses may be delivered, and the IVL catheter can be repositioned within the lesion. For diffuse lesions involving different reference diameters, IVL catheters of different sizes may be utilized.
  Arms: Intensive Preconditioning Group
Device: Routine preconditioning strategy — This includes compliant balloons, non-compliant balloons, cutting/scoring balloons, excimer laser, and rotational atherectomy, to be determined at the operator's discretion
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to investigate whether the clinical outcomes of combined application of intravascular lithotripsy (IVL) following routine preconditioning are superior to those of routine preconditioning alone in patients with moderate-to-severe coronary artery calcification (CAC). Its core research questions are as follows:

A. To evaluate whether routine or combined application of shockwave intravascular lithotripsy can effectively reduce the target vessel failure rate in moderate-to-severe coronary artery calcification lesions.

B. To evaluate the long-term prognosis of patients with coronary artery calcification.

The researchers will compare the experimental group (routine preconditioning plus IVL) and the control group (routine preconditioning alone) to determine whether the combined use of intravascular lithotripsy following routine preconditioning can improve patient prognosis.

DETAILED DESCRIPTION:
Revascularization of severe coronary artery calcification (CAC) lesions is associated with high technical difficulty and poor prognosis, and remains one of the major unmet challenges in the diagnosis and treatment of coronary heart disease (CHD) at present. As an important marker for the severity of atherosclerosis, CAC is closely correlated with the risk of recurrent cardiovascular events after revascularization and future cardiovascular events, with severe CAC lesions increasing the incidence of these events by 20%-40%. Despite existing research on the pathogenesis, progression, risk stratification and therapeutic strategies of CAC, there is a lack of standardized criteria for selecting medical or surgical treatment strategies and optimized revascularization protocols for CAC patients. Therefore, optimizing current revascularization strategies is of great significance.

The proportion of patients with coronary artery calcification (CAC) is on the rise among those undergoing percutaneous coronary intervention (PCI).Existing studies have found that the prevalence of CAC lesions ranges as high as 67% to 90% in the middle-aged and elderly populations. Research indicates that CAC significantly elevates the risk of intraoperative and postoperative complications of PCI, further increasing the likelihood of in-stent restenosis and repeat revascularization, which ultimately leads to a higher risk of mortality. Current preconditioning strategies prior to stent implantation for CAC include high-pressure balloon dilation, cutting balloon dilation, rotational atherectomy, and excimer laser ablation, among other approaches.However, most existing studies have focused on comparing the efficacy of different preconditioning methods-such as the superiority of ultra-high-pressure balloons versus cutting balloons, or rotational atherectomy versus cutting balloons-and have mainly emphasized stent implantation success rates and immediate stent expansion outcomes, while neglecting the long-term prognosis of patients. In particular, relevant research remains insufficient regarding combination therapy regimens that integrate multiple preconditioning methods. In recent years, numerous domestic and international studies have confirmed the efficacy of shockwave balloon technology in the treatment of coronary calcified lesions, which can significantly reduce the rate of stent implantation failure and improve stent expansion rate. Nevertheless, the strategy of intensive preconditioning combined with shockwave balloon therapy still requires verification through large-sample randomized controlled clinical trials.

With population aging and the rising incidence of diabetes mellitus and renal insufficiency, the proportion of patients with CAC lesions is expected to further increase. Therefore, it is particularly important to explore optimized strategies for improving the poor revascularization outcomes in CAC patients.

In summary, by optimizing revascularization strategies, this study aims to establish a more precise and efficient diagnosis and treatment pathway for CAC. Subsequent randomized controlled clinical trials will further clarify the value of these strategies, laying a foundation for promoting breakthroughs in the clinical diagnosis and treatment of cardiovascular diseases, which is of great significance for improving the national cardiovascular health level.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Acute or chronic coronary syndrome requiring PCI
* De novo coronary lesions (excluding bypass grafts and prior stented lesions) with a target vessel reference diameter of ≥ 2.5 mm and ≤ 4.0 mm
* Moderate to severe calcification, meeting one of the following criteria: • Intravascular imaging criteria: IVUS calcium score ≥ 2 points (IVUS scoring standards: a. Calcification > 270 degrees and length > 5 mm; b. Circumferential calcification (360 degrees); c. Calcific nodules; d. Vessel diameter < 3.5 mm) OCT calcium score ≥ 3 points (OCT scoring standards: a. Calcification ≤ 180 degrees: 0 points; > 180 degrees: 2 points; b. Thickness ≤ 0.5 mm: 0 points; > 0.5 mm: 1 point; c. Length ≤ 5 mm: 0 points; > 5 mm: 1 point) • Contrast-based classification criteria apply when intravascular imaging devices cannot pass: Coronary angiography shows clear high-density calcific shadows visible during cardiac pulsation, or clear high-density calcific shadows visible both during and without cardiac pulsation, with the length of calcific shadows on both sides of the target lesion > 5 mm.
* Willing and able to provide written informed consent

Exclusion Criteria:

* Patients under 18 years of age
* Patients unable to provide informed consent
* Pregnant or lactating female patients (pregnancy test must be performed within 7 days before surgery for women of childbearing age)
* Thrombus detected by angiography or intravascular imaging
* Patients with an expected life expectancy of less than 1 year
* Hemodynamically unstable patients
* Patients with known contraindications to heparin, anticoagulants, antiplatelet drugs, contrast agents, or other related medications
* Patients with active bleeding
* Patients with a new-onset stroke or transient ischemic attack (TIA) within 90 days before enrollment
* Patients scheduled to undergo other cardiac interventional procedures or cardiac surgery within 30 days after PCI
* Patients with ST-segment elevation myocardial infarction (STEMI) or cardiogenic shock occurring within 7 days
* Severe renal insufficiency (eGFR ≤ 30 ml/min)
* Left main coronary artery disease
* Presence of type C-F dissection in the target vessel
* Aneurysm within 10 mm of the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1096 (Actual)
Dates: Start 2025-10-24 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
target vessel failure rate | 1month; 12 months; 24 months
  24-month target vessel failure (TVF) rate (a composite endpoint of cardiovascular death, target vessel myocardial infarction [TVMI], and clinically indicated target vessel revascularization [TVR])

SECONDARY OUTCOMES:
MACE | 1 month; 12 months; 24 months
  Including cardiovascular death, myocardial infarction, ischemia-driven revascularization, and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Bingchen Liu, Phd,MD, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China; Bingchen Liu, Phd,MD, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (4):
- China (4):
  - The First Affiliated Hospital of Nanchang University (FAHNU), Nanchang, Jiangxi
  - The People's Hospital of Liaoning Province, Shenyang, Liaoning
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Tianjin Fourth Central Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes